CLINICAL TRIAL: NCT02854462
Title: A Randomised Control Trial to Test the Effect of Parents' Inference-eliciting Questions During Shared Book Reading on 4-year-olds' Listening Comprehension
Brief Title: Supporting Children's School Readiness.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: University of Leeds (Other)
Responsible Party: Principal Investigator, Danielle Matthews, Reader in Cognitive Development, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: R/139470-11-1-INFERENCE
Record Dates: First submitted 2016-07-27; First posted 2016-08-03 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Language Development
Keywords: Language Development; Shared Picture Book reading; Preschoolers; Inference making

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Language comprehension intervention (Experimental): The intervention will run for 4 weeks. Caregivers will be provided with storybooks (e.g., Percy the Park Keeper) that have been amended to include inference-eliciting questions. Caregivers will be trained (with a video) to ask these questions and respond to their children's answers during shared reading sessions. They will be asked to read one book per day. Caregivers will keep a reading diary.
  Interventions: Behavioral: Language comprehension intervention
- Counting intervention (Active Comparator): The intervention will run for 4 weeks. Caregivers will be provided with a book 'At home with counting' that is made up of age appropriate maths exercises. Caregivers will trained (with a video) to work through one page of the book per day. This should take the same amount of time as the activity in the language intervention condition. Caregivers will keep a counting diary.
  Interventions: Behavioral: Counting intervention

INTERVENTIONS:
Behavioral: Language comprehension intervention
  Arms: Language comprehension intervention
Behavioral: Counting intervention
  Arms: Counting intervention

SUMMARY:
The aim of this project is to test whether training parents to ask their children 'inference- eliciting' questions during book reading is effective in promoting story comprehension for 4-year-olds from a range of socio-economic backgrounds.

DETAILED DESCRIPTION:
Language comprehension relies on the ability to make local and global inferences (e.g., inferring what a pronoun refers to, or inferring why a protagonist in a story did something based on information distributed through the text). These skills develop in the preschool years and are demonstrated when children make sense of stories that are read to them. While important for later reading ability and academic success, relatively little is known about whether anything can be done to improve inference-making skills in the preschool years. One possibility is that parent-child book reading would help. During book reading, some parents naturally ask their children questions about the story that would require them to make inferences about the text. The current study is designed to test whether doing this promotes children's ability to make inferences. Half the parents in this study will be given books with inference eliciting questions added to them and will be provided with training about how to ask these questions and respond to their children's answers. The other half of the parents will be given a maths exercise book and asked to spend the same amount of time per day working through this.

ELIGIBILITY:
Inclusion Criteria:

Children are:

First born Full term (i.e. born no more than 3 weeks prematurely) With birth weight over 2.5 kg Being raised as monolingual English speakers

Exclusion Criteria:

Neither caregivers nor infants have any significant known physical, mental or learning disability.

Ages: 50 Months to 56 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
Change after 4 weeks in children's ability to answer inference questions. | Baseline: when child is 4 years 3 months. Post test: 4 weeks post intervention
  An age-appropriate test of inferencing ability has been developed for this study including vignettes developed by the Language and Reading Research Consortium. Children listen to short vignettes and are then asked questions that require them to make local and global inferences based on the information in the stories.

SECONDARY OUTCOMES:
Change in NFER baseline assessment | Baseline: when child is 4 years 3 months - 4 years 6 months. Post test: 4 weeks post intervention
  This is an age appropriate test of maths and language ability.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle E Matthews, PhD, Principal Investigator — University of Sheffield; Catherine Davies, PhD, Principal Investigator — University of Leeds
Locations (1):
- University of Sheffield, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Yes. IPD will be archived in accordance with the guidelines and protocol of the University of Sheffield, the UK Data Archive and the ESRC's Research Data Policy. With parents' permission, data will be made available in a timely manner, after outcomes have been published together with appropriate metadata in line with ESRC policy around data archiving.